CLINICAL TRIAL: NCT05217316
Title: Assess the Impact of Virtual Supervised Tooth Brushing on Dental Caries and Quality of Life Among Primary School Children in Riyadh, KSA
Brief Title: Impact of Virtual Supervised Tooth Brushing Among Primary School Children in Riyadh, KSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-21-5925
Record Dates: First submitted 2021-12-14; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Dental Caries in Children
Keywords: Toothbrushing; Quality of Life

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial comparing virtual supervised tooth brushing program against conventional oral hygiene program (lecture and tooth brushing demonstration). 1280 children in 20 primary schools in Riyadh, Saudi Arabia will be recruited to the trail. Schools are the unit of clustering. Schools will be randomly selected and allocated in two groups, intervention, and control group (10 schools for each group). Clinical assessment for dental caries will be conducted in four points (baseline, 6 months, 12 months, 18 months). Both groups will receive oral assessment and both will receive a videos five times a week that illustrate a unified toothbrushing technique and remind the child to brush their teeth. The intervention lies in which the intervention group will receive a supervised virtual toothbrushing performed once a week for each child.
Who Masked: Investigator
Masking Description: 20 primary schools in Riyadh, Saudi Arabia will be recruited to the trail. Schools are the unit of clustering will be randomly selected and allocated to groups. The schools who did not respond and refused to participate will be dropped and replaced randomly from the selected list. All data entry and management will be carried out by the study principal investigator. This will be applied by pseudo-anonymization, an artificial identifier (code) will be assigned to each subject as he enrolled in the study. All the study team members will deal with coded data while collecting or analyzing information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group will receive a videos five times a week that illustrate a unified toothbrushing technique and remind the child to brush their teeth.
- Intervention Group (Experimental): Both groups will receive a videos five times a week that illustrate a unified toothbrushing technique and remind the child to brush their teeth. The intervention lies in which the intervention group will receive a supervised virtual toothbrushing performed once a week for all students by dental hygienist that will be performed through a prescheduled virtual appointment for each child.
  Interventions: Behavioral: Supervised Virtual Toothbrushing

INTERVENTIONS:
Behavioral: Supervised Virtual Toothbrushing — A supervised virtual toothbrushing performed once a week for all students by dental hygienist that will be performed through a prescheduled virtual appointment for each child. All virtual appointments will be conducted using the collaboration of two national platforms. "Mawid", a Ministry of health (MOH) Central Appointment System, to be used by the subjects. And "ANAT" system, a Saudi Commission for Health Specialists (SCHS) application for the hygienists to use for their virtual supervision.
  Arms: Intervention Group

SUMMARY:
Dental caries is one of the most common diseases affecting children in Saudi Arabia despite the availability of free dental services. The combination of the large burden of untreated caries among school children, low uptake of dental services when asymptomatic and the availability of free dental services makes Saudi Arabia a unique setting for school-based dental programs. Despite the availability of free dental services provided through the Ministry of Health, universities' hospitals and health services of the Ministry of Defense, most Saudis visit the dentist only when in pain.

As schools are carried out virtually and Saudi Arabia has proved effective IT infrastructure, virtual supervised tooth brushing is a proposed initiative. It is also an opportunity for targeting a large portion of the population with a high level of disease as a quarter of the Saudi population is younger than 15 years.

DETAILED DESCRIPTION:
Background Dental caries is one of the most common diseases that afflict children in the Kingdom of Saudi Arabia and despite the availability of free dental services provided through the Ministry of Health, universities, hospitals and health services of the Ministry of Defense, most Saudis visit the dentist only when they are in pain thus, they reach the health care when they need complex care.

Aim The aim is to assess the impact of virtual supervised toothbrushing on dental caries and quality of life among primary school children in Riyadh, KSA.

Research Methodology This is a cluster randomized controlled trial comparing virtual supervised tooth brushing program against conventional oral hygiene program (lecture and tooth brushing demonstration). A 1280 children in 20 primary schools in Riyadh, Saudi Arabia will be recruited to the trail. Schools are the unit of clustering will be randomly selected and allocated to groups. Clinical assessment for dental caries will be conducted in four points (baseline, 6 months, 12 months, 18 months) by dental hygienist using World Health Organization criteria. Data on socio-demographic behavioral factors and children's quality of life will be collected at baseline and 12 months later through a structured questionnaire. The primary outcome is the change in the number of teeth with untreated dental caries in both primary and permanent teeth over 18 months. The secondary outcomes are the change in the frequency of brushing per day and the impact of oral health on the child's daily life (QoL).

Research Significance Schools are carried out virtually and Saudi Arabia has proved effective IT infrastructure, virtual supervised tooth brushing is a proposed initiative. It is also an opportunity for targeting a large portion of the population with a high level of disease as a quarter of the Saudi population is younger than 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 9 years (4th grade at school) at baseline
* Both Saudis and non-Saudis
* Children for whom the person with parental responsibility has signed the consent form

Exclusion Criteria:

* Children in 5th and 6th grade (11- 12-year-olds) as they would have left schools by the time of the follow-up assessment (18 months later).
* Children who refuse to participate in the study

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1280 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dental Caries | 18 months
  The study primary outcome is the change in the number of teeth with untreated dental caries in both primary and permanent teeth over 18 months.

SECONDARY OUTCOMES:
Frequency of Brushing | 1 year
  The change in the frequency of brushing per day
Quality of Child's Daily Life | 18 months
  The impact of oral health on the child's daily life (QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Haya Alayadi, PhD, Principal Investigator — King Saud University
Locations (1):
- Haya Alayadi, Riyāḑ, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
This will be applied by pseudo-anonymization. A separate file all personal identifiable information for all subjects will be kept in a separate file by the principal investigator. In addition, an artificial identifier (code) will be assigned to each subject as he enrolled in the study. All the study team members will deal with coded data while collecting or analyzing information.
  Only the codes will be used in data entry without any identifiable personal information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2 years
Access Criteria: Only the authorized team members will grant access to the study data.

REFERENCES:
- [Background] Almas K, Al-Malik TM, Al-Shehri MA, Skaug N. The knowledge and practices of oral hygiene methods and attendance pattern among school teachers in Riyadh, Saudi Arabia. Saudi Med J. 2003 Oct;24(10):1087-91. PMID 14578974
- [Background] El Bcheraoui C, Tuffaha M, Daoud F, Kravitz H, AlMazroa MA, Al Saeedi M, Memish ZA, Basulaiman M, Al Rabeeah AA, Mokdad AH. Use of dental clinics and oral hygiene practices in the Kingdom of Saudi Arabia, 2013. Int Dent J. 2016 Apr;66(2):99-104. doi: 10.1111/idj.12210. Epub 2016 Jan 7. PMID 26749526
- [Background] Al-Yousuf M, Akerele TM, Al-Mazrou YY. Organization of the Saudi health system. East Mediterr Health J. 2002 Jul-Sep;8(4-5):645-53. PMID 15603048
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of untreated caries: a systematic review and metaregression. J Dent Res. 2015 May;94(5):650-8. doi: 10.1177/0022034515573272. Epub 2015 Mar 4. PMID 25740856
- [Background] Kassebaum NJ, Smith AGC, Bernabe E, Fleming TD, Reynolds AE, Vos T, Murray CJL, Marcenes W; GBD 2015 Oral Health Collaborators. Global, Regional, and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries, and Risk Factors. J Dent Res. 2017 Apr;96(4):380-387. doi: 10.1177/0022034517693566. PMID 28792274
- [Background] Holland WW, Stewart S. Screening in health care. Benefit or bane? London: The Nuffield Provincial Hospitals Trust; 1990.
- [Background] World Health Organization. Oral health surveys: basic methods. 5th ed. Geneva: World Health Organization; 2013.
- [Derived] Alayadi H, Alsiwat A, AlAkeel H, Alaskar M, Alwadi M, Sabbah W. Impact of virtual supervised tooth brushing on caries experience and quality of life among primary school children: study protocol for a randomized controlled trial. Trials. 2023 Feb 20;24(1):118. doi: 10.1186/s13063-023-07111-8. PMID 36803406